CLINICAL TRIAL: NCT01962714
Title: A Trial of Loving-Kindness Meditation and Cognitive Processing Therapy for PTSD
Brief Title: Loving-Kindness Meditation for PTSD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MHBA-006-13S; 5I01CX000857-02 (NIH)
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Results first posted 2020-02-27 (Actual); Last update posted 2020-03-17 (Actual); Status verified 2020-03

CONDITIONS: Posttraumatic Stress Disorder; Depression
Keywords: Behavior therapies, cognitive; Mindfulness; Emotion; Group therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Loving-Kindness Meditation (Experimental): A 12-week duration, 90-minute per session Loving-Kindness Meditation (LKM) course, taught in groups of 10 participants.
  Interventions: Behavioral: Loving-Kindness Meditation
- Cognitive Processing Therapy - Cognitive Only (Active Comparator): A 12-week duration, 90-minute per session Cognitive Processing Therapy (CPT) course, taught in groups of 10 participants.
  Interventions: Behavioral: Cognitive Processing Therapy

INTERVENTIONS:
Behavioral: Loving-Kindness Meditation — 12-week loving-kindness meditation course
  Arms: Loving-Kindness Meditation
Behavioral: Cognitive Processing Therapy — 12-week CPT course
  Arms: Cognitive Processing Therapy - Cognitive Only

SUMMARY:
This randomized controlled trial will assess whether a novel complementary and alternative medicines (CAM) intervention, Loving-kindness Meditation (LKM), is not meaningfully inferior to another group-based PTSD treatment , Cognitive Processing Therapy (Cognitive Only version; CPT-C) for reductions in PTSD and depressive symptoms. 170 male and female Veterans with current PTSD will be randomized to LKM or CPT-C. The investigators hypothesize that Veterans randomized to LKM will report mean reductions in PTSD and depressive symptom severity that are not meaningfully worse than CPT-C. The investigators further hypothesize that reductions in posttraumatic maladaptive beliefs will more strongly mediate PTSD and depressive symptom improvement for those assigned to CPT-C than those assigned to LKM.

DETAILED DESCRIPTION:
Aim 1: Evaluate if LKM is non-inferior to CPT-C in producing reductions in PTSD symptoms among Veterans with current PTSD. Aim 2: Evaluate the non-inferiority of LKM and CPT-C in producing reductions in depressive symptoms among Veterans with current PTSD. Exploratory Aim: Evaluate potential mediators of response to LKM and to CPT to provide preliminary information regarding whether they are consistent with the mechanisms of change conceptualized by each intervention to be associated with improvement in PTSD and depression.

Methods: A randomized controlled non-inferiority trial comparing LKM to CPT-C. In the proposed project 170 Veterans with PTSD will be randomized to LKM or CPT-C. Comprehensive assessments will be performed at baseline as well as at the end of the 12-week interventions and 3 and 6 months later. PTSD symptoms, depression, posttraumatic maladaptive cognitions and self-compassion will be assessed weekly during the treatment phase to assess temporality of change and to assess mediators of outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Current Diagnostic and Statistical Manual of Mental Disorder (DSM)-5 diagnosis of PTSD,
* 18 or over,
* English fluency,
* Willingness to not participate in Mindfulness-Based Stress Reduction or other meditation programs, as well as Prolonged Exposure (PE) or CPT during the study period.

Exclusion Criteria:

* Any of the following substance use criteria: 1) Use in the past 90 days of illicit substance (do not include cannabis)/ street drug (non-prescribed); 2) Use in the past 90 days of prescription drug of abuse, use is not as prescribed AND poses safety concern
* Alcohol involvement that poses a safety concern or is associated with inability to follow through on assessments and class attendance as evinced by current drinking AND dt's or seizure in past year
* Suicidal or homicidal ideation with intent or plan
* Attempted harm to Self or others in the past month
* A lifetime psychotic disorder or current psychotic symptoms
* Uncontrolled bipolar disorder (ie current mania, current hypomania is not an exclusion)
* Chart diagnoses of borderline personality disorder or antisocial personality disorder
* In-patient admission for psychiatric reasons within the past month
* Prior participation in LKM or CPT
* Dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2014-12-01 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2018-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J. Kearney, MD, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
A de-identified, anonymized dataset will be created and shared.

REFERENCES:
- [Result] Kearney DJ, Malte CA, McManus C, Martinez ME, Felleman B, Simpson TL. Loving-kindness meditation for posttraumatic stress disorder: a pilot study. J Trauma Stress. 2013 Aug;26(4):426-34. doi: 10.1002/jts.21832. Epub 2013 Jul 25. PMID 23893519
- [Derived] Kearney DJ, Malte CA, Storms M, Simpson TL. Loving-Kindness Meditation vs Cognitive Processing Therapy for Posttraumatic Stress Disorder Among Veterans: A Randomized Clinical Trial. JAMA Netw Open. 2021 Apr 1;4(4):e216604. doi: 10.1001/jamanetworkopen.2021.6604. PMID 33861329

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Loving-Kindness Meditation | Cognitive Processing Therapy - Cognitive Only
Started | 91 | 93
Immediate Post-treatment Assessment | 63 | 57
3-month Follow-up | 58 | 56
Completed | 61 | 60
Not Completed | 30 | 33

BASELINE CHARACTERISTICS:
Groups:
- Loving-Kindness Meditation: The intervention consisted of 12 weekly 90-minute group sessions. In Loving-Kindness Meditation, a person sits and calls to mind a particular person (e.g., a good friend) and silently repeats phrases that invoke goodwill for that person, e.g., the desire for safety, happiness, health, and peace. Over 12 weeks, the practice expands to bring to mind other individuals or categories of people, including themselves, neutral persons, and those who have caused difficulty or harm, changing the phrases as needed. Participants are asked to notice any thoughts and feelings elicited by the phrases with an attitude of kindness, curiosity, and non-judgment, regardless of content. Each session begins with either mindfulness meditation (weeks 1 & 2) or LKM meditation (weeks 3 through 12) followed by group discussion and additional LKM teaching and practice. Homework for LKM consisted of 30 minutes of meditation 6 days per week using compact disks (CDs) as well as informal LKM practice in daily life.
- Cognitive Processing Therapy - Cognitive Only: CPT-C does not include writing a trauma narrative. The intervention is based on Resick and colleagues' manual for treating PTSD among military veterans, which combines cognitive restructuring with emotional processing of trauma- related content. Sessions initially focus on rigid or inaccurate beliefs about the traumatic event itself, which often reflect self-blame or hindsight bias. Later sessions address over-generalized beliefs about self and others that result from a traumatic event relevant to five key areas: safety, trust, power, esteem, and intimacy. Clients learn to identify and modify their beliefs to develop more balanced, flexible, and ultimately, more adaptive beliefs. Homework for CPT-C consisted of 30 minutes of homework 6 days a week, including writing an impact statement at the beginning and the end of treatment and completing worksheets and exercises regarding safety, trust, power/control, esteem, and intimacy.
- Total: Total of all reporting groups
Arm/Group | Loving-Kindness Meditation | Cognitive Processing Therapy - Cognitive Only | Total
Number analyzed (Participants) | 91 | 93 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (12.5) | 56.1 (13.7) | 57.1 (13.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Male | 77 | 76 | 153
  Gender: Female | 13 | 17 | 30
  Gender: Transgender | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 88 | 87 | 175
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 3 | 3
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 20 | 44
  White | 53 | 54 | 107
  More than one race | 11 | 12 | 23
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 91 | 93 | 184
Clinician-Administered PTSD Scale for Diagnostic and Statistical Manual (DSM)-5 (CAPS-5) [Mean (Standard Deviation); unit: units on a scale] — The CAPS-5 structured interview was performed by a clinician blinded to randomization arm. Range 0-80; higher scores indicate worse PTSD.
  units on a scale | 35.54 (12.12) | 35.53 (11.48) | 35.53 (11.77)

OUTCOME MEASURES:

1. Primary Outcome: Clinician Administered PTSD Scale (CAPS-5) Score
Description: PTSD diagnostic severity was measured using the 30-item CAPS-5 structured interview (range 0-80; higher scores indicate worse PTSD). Linear mixed effects models (LMM) were used to analyze continuous outcomes, with time and time by treatment interaction included as fixed effects to determine if differences exist between conditions by time. Non-inferiority of LKM to CPT-C was claimed if the lower limit of the 95% confidence interval for difference in change rate from baseline to 6-month follow-up in mean CAPS or depression score was greater than (i.e., did not extend beyond) negative delta (defined as 5 points on the CAPS-5 measure). A 2-sided 95% confidence interval of the difference in change rate from baseline to 6-month follow-up between groups (CPT-C minus LKM) was calculated, with a positive value indicating a greater reduction in scores from baseline for LKM compared to CPT-C.
Time Frame: 6 months post-intervention
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Loving-Kindness Meditation | Cognitive Processing Therapy - Cognitive Only
Number analyzed (Participants) | 91 | 93
units on a scale | 25.92 [22.62 to 29.23] | 28.02 [24.72 to 31.32]
Statistical Analysis 1: Comparison: Loving-Kindness Meditation vs Cognitive Processing Therapy - Cognitive Only; The non-inferiority of LKM with respect to CPT-C was analyzed using the 95% confidence interval for the group x time interaction term, with non-inferiority of LKM to CPT-C claimed if the lower limit of the 95% confidence interval was greater than (i.e., did not extend beyond) negative delta; Test type: Non-Inferiority — The primary outcome of non-inferiority of LKM relative to CPT-C was assessed using a non-inferiority margin of 5 points on the CAPS-5, which represents 0.5 SD of baseline PTSD symptoms based on data indicating the SD of baseline CAPS-5 scores is approximately 10 in a large sample (N=198) of treatment-seeking veterans; Mean Difference (Final Values) = 2.09, 95% CI 2-sided [-2.59 to 6.78] — Non-inferiority of LKM to CPT-C was analyzed as the change rate from baseline to 6-month follow-up between groups (CPT-C minus LKM), with a positive value indicating a greater reduction in scores for LKM compared to CPT-C

2. Primary Outcome: NIH Patient-Reported Outcomes Measurement Information System (PROMIS) Depression Score
Description: Depression was assessed using the National Institute of Health (NIH) Patient-Reported Outcomes Measurement Information System (PROMIS) depression measure. This scale utilizes item-response theory and is scored using a T-score metric with a mean of 50 and SD=10 in the US general population. Higher scores indicate more severe depression.
Time Frame: 6 months post-intervention
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Loving-Kindness Meditation | Cognitive Processing Therapy - Cognitive Only
Number analyzed (Participants) | 91 | 93
units on a scale | 58.88 [56.86 to 60.91] | 61.22 [59.21 to 68.23]
Statistical Analysis 1: Comparison: Loving-Kindness Meditation vs Cognitive Processing Therapy - Cognitive Only; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — For depression, the non-inferiority margin was 4 points on the PROMIS depression measure, which has been defined as the minimally important difference and corresponds to a Cohen's d effect size of approximately 0.50; Mean Difference (Final Values) = 2.34, 95% CI 2-sided [-0.52 to 5.20] — Non-inferiority of LKM with respect to CPT-C was analyzed as the change rate from baseline to 6-month follow-up between groups (CPT-C minus LKM), with a positive value indicating a greater reduction in scores from baseline for LKM compared to CPT-C

ADVERSE EVENTS:
Time Frame: From baseline to 6-month follow-up (approximately 9 months total).
Description: We prospectively monitored hospitalizations, suicidality and death. In addition we recorded events according to the following criteria: An increase of 20 or more points on the total CAPS-5 score since the last assessment point or an increase in depression severity of 2 or more severity categories using a rubric that transformed PROMIS depression values scores to Patient Health Questionnaire (PHQ)-9 scores and categories
Arm/Group | Loving-Kindness Meditation | Cognitive Processing Therapy - Cognitive Only
All-Cause Mortality (participants affected / at risk) | 2/91 | 0/93
Serious Adverse Events (participants affected / at risk) | 5/91 | 3/93
Other Adverse Events (participants affected / at risk) | 11/91 | 18/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loving-Kindness Meditation (N=91) | Cognitive Processing Therapy - Cognitive Only (N=93)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Inpatient psychiatric admission (Psychiatric disorders) | 1 (1) | 0 (0)
Risk of Harm to Others (Psychiatric disorders) | 0 (0) | 1 (1)
Suicidality with Intent or Plan requiring staff intervention (Psychiatric disorders) | 4 (4) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Loving-Kindness Meditation (N=91) | Cognitive Processing Therapy - Cognitive Only (N=93)
Increase in depression score (Psychiatric disorders) | 7 (91) | 14 (93) — An increase in depression severity of 2 or more severity categories was categorized as an adverse event (AE). A rubric was utilized that transformed PROMIS depression scores to PHQ-9 scores for this purpose.
Increase in PTSD severity score (Psychiatric disorders) | 4 (91) | 3 (93) — An increase of 20 or more points on the CAPS-5 score since the last assessment was categorized as an AE.
Risk of harm to others (Psychiatric disorders) | 0 (0) | 1 (93)

LIMITATIONS AND CAVEATS:
The study involved predominantly male veterans from one facility; the results may not generalize to nonveterans or veterans in other regions. Treatment credibility and adequacy of blinding of the clinician-assessor of PTSD symptoms were not assessed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-31): https://cdn.clinicaltrials.gov/large-docs/14/NCT01962714/Prot_SAP_000.pdf